CLINICAL TRIAL: NCT00496483
Title: A Phase II, Open-Label, Multi-Center Prospective, Conversion Study in Stable Kidney Transplant Patients to Compare the Pharmacokinetics of LCP-Tacro Tablets Once-A-Day to Prograf® Capsules Twice-A-Day
Brief Title: Pharmacokinetics of LCP-Tacro in Stable Kidney Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCP-Tacro 2011
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Renal Failure
Keywords: Tacrolimus; Pharmacokinetics; Kidney Transplantation
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LCP-Tacro (tacrolimus) (Active Comparator): Experimental: LCP Tacro; investigational product LCP-Tacro tablets were provided in 3 strengths: 1 mg, 2 mg, and 5 mg oral tablets.
  Interventions: Drug: LCP Tacro (tacrolimus); Drug: Prograf

INTERVENTIONS:
Drug: LCP Tacro (tacrolimus) — Prograf will be administrated twice a day, per product labeling, with an interval of 12 ± 1 hours between the morning and evening doses. Patients will continue on the same dose on Day0 through Day 7 to maintain target trough levels of 7-12 ng/mL. On the morning of Day 8, following the final blood draw for the PK assessment, patient will be converted to LCP-Tacro using the conversion Ratio 0.66-0.8. LCP-Tacro tablets will be administered orally once daily in the morning, with an interval of 24 ± 1 hours between doses.
  Other Names:
  Tacrolimus modified-release LCP-Tacro tablets were provided in 3 strengths: 1 mg, 2 mg, and 5 mg oral tablets.
  Other Names: tacrolimus
Drug: Prograf — Prograf will be administrated twice a day, per product labeling, with an interval of 12 ± 1 hours between the morning and evening doses. Patients will continue on the same dose on Day0 through Day 7 to maintain target trough levels of 7-12 ng/mL. On the morning of Day 8, following the final blood draw for the PK assessment, patient will be converted to LCP-Tacro using the conversion Ratio 0.66-0.8. LCP-Tacro tablets will be administered orally once daily in the morning, with an interval of 24 ± 1 hours between doses.
  Other Names:
  Tacrolimus modified-release LCP-Tacro tablets were provided in 3 strengths: 1 mg, 2 mg, and 5 mg oral tablets.
  Other Names: Tacrolimus

SUMMARY:
A three sequence, open-label, multi-center, prospective, study in stable kidney transplant patients to assess and compare the pharmacokinetics (Cmax, C24, and AUC), and safety of LCP-Tacro (tacrolimus) tablets versus Prograf (tacrolimus) capsules.

DETAILED DESCRIPTION:
A three sequence, open-label, multi-center, prospective, study in stable kidney transplant patients to assess and compare the pharmacokinetics (Cmax, C24, and AUC), and safety of LCP-Tacro (tacrolimus) tablets versus Prograf (tacrolimus) capsules.

Stable kidney transplant patients who fulfill all I/E criteria will be enrolled and kept on Prograf for 7 days. Following a 24-hour PK study on Day 7 to determine pharmacokinetics for Prograf, all patients will be converted to once daily LCP-Tacro for 7 days with no dose changes allowed. On Day 14 and Day 21 a 24-hour LCP-Tacro PK study will be performed. On Day 22 patients will be converted back to their original twice daily dose of Prograf for a safety follow-up period of 30 days ending with a safety assessment on day 53.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years of age who are recipients of a renal transplant at least 6 months prior to enrollment
* Patients on oral Prograf therapy as part of their maintenance immunosuppression therapy, with stable doses and trough levels of tacrolimus of 7-12 ng/mL for at least two weeks prior to enrollment.
* Patients maintained on concurrent immunosuppression with mycophenolate mofetil (MMF, CellCept) or mycophenolic acid delayed-release tablets (Myfortic), with stable doses for at least two weeks prior to enrollment
* Patients with serum creatinine < 2.0mg/dL prior to enrollment
* Able to swallow study medication
* Patients capable of understanding the purposes and risks of the study, who can give written informed consent and who are willing to participate in and comply with the study
* Women of childbearing potential must have a negative serum pregnancy test within seven days prior to receiving study medication
* Patients who successfully pass a drug screen

Exclusion Criteria:

* Recipients of any transplanted organ other than a kidney
* White blood cell count < 2.8 x 10^9 /L
* Patients who are receiving a total dose of Prograf for 24 hours < 3mg
* Patients unable or unwilling to provide informed consent
* Pregnant or nursing women
* Patients with reproductive potential who are unwilling/unable to use a double barrier method of contraception
* Administration of other investigational agent in the three months prior to enrollment
* Patient receiving any drug interfering with tacrolimus metabolism
* Patients who have taken sirolimus within the past three months prior to screening
* Patient with an episode of acute cellular requiring antibody therapy within the 6 months prior to enrollment
* Patient treated for acute cellular rejection within the 30 days prior to enrollment
* Patient who is HCV negative and has received an HCV positive (HCV RNA by PCR or HCV antibody) donor kidney
* Patient has a current malignancy or a history of malignancy (within the past 5 years), except basal or non-metastatic squamous cell carcinoma of the skin that has been treated successfully
* Patient has uncontrolled concomitant infection, a systemic infection requiring treatment, or any other unstable medical condition that could interfere with the study objectives
* Patient has severe diarrhea, vomiting, active peptic ulcer or gastrointestinal disorder that may affect the absorption of tacrolimus
* Patient will require therapy with any immunosuppressive agent other than those prescribed in the study
* Patient has a known hypersensitivity to corticosteroids, mycophenolate mofetil, mycophenolic acid or tacrolimus
* Patient has any form of current substance abuse, psychiatric disorder or a condition that, in the opinion of the Investigator, may invalidate communication with the Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Glicklich, MD, Study Director — Veloxis Pharmaceuticals
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - Methodist Hospital Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- LCP-Tacro: All Patients received Prograf for 7 days, then all patients were converted to once daily LCP-Tacro for 14 days. One dose adjustment up or down 25% was permitted on Day 15.
  On Day 22 patients were converted back to their original twice daily dose of Prograf for a safety follow-up period of 30 days.
  LCP-Tacro 1 mg, 2 mg and 5 mg tablets administered orally QD, dosing per conversion algorithm to maintain tacrolimus trough concentrations between 7 to 12 ng/mL.
Period: Overall Study
Arm/Group | LCP-Tacro
Started | 60
Dosed | 51
Completed | 48
Not Completed | 12
Not completed — Not dosed | 9
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Groups:
- LCP-Tacro: LCP-Tacro 1 mg, 2 mg and 5 mg tablets administered orally QD, dosing per conversion algorithm to maintain tacrolimus trough concentrations between 7 to 12 ng/mL.
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Secondary Outcome: Tacrolimus Pharmacokinetics (Cmax and Cavg) Was Measured at Day 21.
Description: Cmax and Cavg was measured at day 21 (Cmin was measured as part of the primary outcome).
Time Frame: 21 days
Population: 48 completed treatment with LCP-Tacro but one patient was excluded from the PP analysis due to inappropriate conversion rate. Another patient discontinued before the Day 21 visit.
  The arithmetic mean and standard deviation is given.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 46
ng/mL
  Cmax | 13.94 (5.84)
  Cavg | 9.08 (2.84)

2. Secondary Outcome: Tacrolimus Pharmacokinetics (Tmax) Was Measured at Day 21.
Description: Tmax was measured at day 21 (Cmin was measured as part of the primary outcome).
Time Frame: 21 days
Population: 48 completed treatment with LCP-Tacro but one patient was excluded from the PP analysis due to inappropriate conversion rate. Another patient discontinued before the Day 21 visit.
Measure: Mean (Full Range); unit: hour
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 46
hour | 6.00 [1.50 to 16.00]

3. Secondary Outcome: Tacrolimus Pharmacokinetics (Fluctuation and Swing) Was Measured at Day 21.
Description: Degree og fluctuation and degree of swing was measured at day 21 (Cmin was measured as part of the primary outcome).
Time Frame: 21 days
Population: 48 completed treatment with LCP-Tacro but one patient was excluded from the PP analysis due to inappropriate conversion rate. Another patient discontinued before the Day 21 visit.
  Arithmetic mean and standard deviation is given below.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 46
percentage
  Fluctuation | 77.04 (50.59)
  Swing | 110.07 (89.23)

4. Primary Outcome: Evaluation of Steady State Tacrolimus Trough Levels (C24).
Description: Patients had a baseline trough level (C24) measured at day 7 before conversion to LCP-Tacro.
Time Frame: 7 days
Population: 48 completed treatment with LCP-Tacro but one patient was excluded from the PP analysis due to inappropriate conversion rate.
  The arithmetic mean and standard deviation is given.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Prograf: Prograf 0.5 mg, 1 mg and 5 mg capsules administered orally twice daily, dosing per conversion algorithm to maintain tacrolimus trough concentrations between 7 to 12 ng/mL.
Arm/Group | Prograf
Number analyzed (Participants) | 47
ng/mL | 7.00 (1.54)

5. Primary Outcome: Evaluation of Steady State Tacrolimus Exposure (AUC 0-24).
Description: Patients had a baseline AUC measured (0 to 24 hours) at day 7 before conversion to LCP-Tacro.
Time Frame: 7 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Prograf: Prograf 0.5 mg, 1 mg and 5 mg capsules administered orally QD, dosing per conversion algorithm to maintain tacrolimus trough concentrations between 7 to 12 ng/mL.
Arm/Group | Prograf
Number analyzed (Participants) | 47
ng*hr/mL | 218.82 (55.99)

6. Primary Outcome: Evaluation of Steady State Tacrolimus Exposure Trough Levels (C24).
Description: Patients were converted from Prograf to LCP-Tacro on day 7. On day 21, a trough level (C24) was measured.
Time Frame: 21 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 46
ng/mL | 6.94 (2.20)

7. Primary Outcome: Evaluation of Steady State Tacrolimus Exposure (AUC 0-24).
Description: Patients were converted from Prograf to LCP-Tacro on day 7. On day 21, AUC was measured (0 to 24 hours).
Time Frame: 21 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 46
ng*hr/mL | 218.03 (68.23)

8. Secondary Outcome: Tacrolimus Pharmacokinetics (Cmax and Cavg) Was Measured at Day 7.
Description: Cmax and Cavg was measured at baseline day 7 (Cmin was measured as part of the primary outcome).
Time Frame: 7 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Prograf
Number analyzed (Participants) | 47
ng/mL
  Cmax | 19.14 (8.15)
  Cavg | 9.12 (2.33)

9. Secondary Outcome: Tacrolimus Pharmacokinetics (Tmax) Was Measured at Day 7.
Description: Tmax was measured at baseline day 7 (Cmin was measured as part of the primary outcome).
Time Frame: 7 days
Population: as for outcome 2
Measure: Mean (Full Range); unit: hour
Arm/Group | Prograf
Number analyzed (Participants) | 46
hour | 1.82 [0.50 to 24.00]

10. Secondary Outcome: Tacrolimus Pharmacokinetics (Fluctuation and Swing) Was Measured at Day 7.
Description: Degree og fluctuation and degree of swing was measured as baseline at day 7 (Cmin was measured as part of the primary outcome).
Time Frame: 7 days
Population: 48 completed treatment with LCP-Tacro but one patient was excluded from the PP analysis due to inappropriate conversion rate.
  Arithmetic mean and standard deviation is given below.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Prograf
Number analyzed (Participants) | 47
percentage
  Fluctuation | 127.41 (57.28)
  Swing | 174.55 (93.72)

11. Secondary Outcome: Safety Evaluation
Description: A combination of deaths, graft failure and biopsy proven acute rejections (BPAR) was used to evaluate the safety.
Time Frame: 52 days
Population: All enrolled patients are included in the safety population.
Measure: Number; unit: participants
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 60
participants
  Death | 0
  Graft failure | 0
  BPAR | 0

ADVERSE EVENTS:
Groups:
- LCP-Tacro: LCP-Tacro 1 mg, 2 mg and 5 mg tablets administered orally QD, dosing per conversion algorithm to maintain tacrolimus trough concentrations between 7 to 12 ng/mL.
  60 patients were enrolled into the study, but only 51 were dosed with LCP-Tacro.
- Prograf: Prograf 0.5 mg, 1 mg and 5 mg capsules administered orally twice daily, dosing per conversion algorithm to maintain tacrolimus trough concentrations between 7 to 12 ng/mL.
  60 patients were entrolled into the study and one withdrew consent right after screening. Therefore 59 patients are inlcuded in the ITT safety set.
Arm/Group | LCP-Tacro | Prograf
Serious Adverse Events (participants affected / at risk) | 2/51 | 0/59
Other Adverse Events (participants affected / at risk) | 35/51 | 19/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=51) | Prograf (N=59)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=51) | Prograf (N=59)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Urinary casts (Investigations) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Dsypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Application site irritation (General disorders) | 1 (1) | 0 (0)
Conjunctuvitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Poor venous access (Vascular disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Immunosuppressant drug level increased (Investigations) | 0 (0) | 1 (1)
Gatroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study is a multicenter collaborative investigation and the clinical trial results are to be published as a collaborative manuscript. Authorship will reflect varying levels of individual contribution to the study by the individual PI's.